CLINICAL TRIAL: NCT06462248
Title: A Single Arm, Open-labelled Phase II Clinical Trial of Anti-CD19 Chimeric Antigen Receptor Modified T-cell (CAR-T) for Treatment of B-cell Haematological Malignancies
Brief Title: Anti-CD19 Chimeric Antigen Receptor Modified T-cell (CAR-T) Therapy for Treatment of B-cell Hematological Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chi Kong Li (Other)
Collaborators: Hong Kong Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Chi Kong Li, Research Professor, Prince of Wales Hospital, Shatin, Hong Kong
Organization: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CU2022
Record Dates: First submitted 2024-06-07; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Lymphoma, Nonhodgkin; Leukemia, Lymphocytic
Keywords: relapsed leukemia; relapsed B-cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphoid; Leukemia; Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: single arm prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Single arm open labelled phase 2 study
  Interventions: Drug: CUCART19

INTERVENTIONS:
Drug: CUCART19 — anti-CD19 chimeric antigen receptor modified T-cell (CAR-T)
  Other Names: anti-CD19 CAR-T

SUMMARY:
CAR-T therapy is now available as a commercial product for treatment of relapsed /refractory acute lymphoblastic leukaemia and B-lymphoma. There is limited access to this new treatment as the product is very expensive. It is imperative to develop cost effective, closed circuit manufacturing systems for CAR-T cells to make CAR-T cells a point-of care production option. Hong Kong Institute of Biotechnology has established a certified GMP facility and utilize the Prodigy system to manufacture CAR-T cells for clinical application. Prince of Wales Hospital and Hong Kong Children's Hospital will conduct the phase II clinical trial to confirm the efficacy and safety of local manufactured CAR-T cell product.

DETAILED DESCRIPTION:
This is a pilot study of CD19 specific CAR-T cells produced by the CliniMACS prodigy system in treatment of paediatric and adult with relapsed or refractory Acute Lymphoblastic Leukemia (ALL) or B cell Non-Hodgkin Lymphoma (NHL).

Our study aims to evaluate the safety and effectiveness of CD19 specific CAR-T cells produced by a closed circuit, point of care, manufacturing system to develop safe and effective CD19 specific CART cells for treatment of relapsed B cell NHL and relapsed refractory B cell ALL in children and adults. The CliniMACS plus system of Miltenyi Biotec is an automated cell separator with proven clinical efficacy. The CliniMACS prodigy system has been successfully used to generate a CD19 CAR T using lentiviral transduction with good efficiency of transduction and the activity of the CAR T cells.

This pilot study using anti-CD19 CAR-T cells generated by the CliniMACS prodigy system will be undertaken in the Prince of Wales Hospital under the Department of Clinical Oncology, Department of Medicine, and the Department of Anatomical & Cellular Pathology. Children will be managed at Hong Kong Children's Hospital. The subjects will comprise of paediatric and adult B cell ALL patients and cohort B of paediatric and adult B cell NHL patients.

Eligible patients will go through Lymphapheresis procedures through central venous access. The cells will then be transferred to the CliniMACS prodigy system where they will be enriched and activated using the transAct CD3/CD28 Kit and transduced with a self-inactivating lentiviral vector encoding a CAR specific for CD19. The cells will be cultured, expanded and tested for efficiency of transduction, sterility and phenotype before preparation for patient use. The CAR-T cell treatment plan is consisted of a course of conditioning chemotherapy, followed by a single infusion of anti-CD19 CAR T cells after completion of conditioning / lymphodepletion chemotherapy. Patients will be observed as an inpatient for 7 days post treatment. Clinical status and progress of the patients, vital signs, blood counts, and blood chemistries will be monitored during and after CAR-T cell therapy. Occurrence of adverse events and serious adverse events will be recorded and managed with standard guidelines. Patients should be regularly followed up for at least two years after CAR T therapy. It is preferably to have long term follow-up of the patients beyond two years to look for any late complications

ELIGIBILITY:
Inclusion Criteria:

Acute Lymphoblastic Leukaemia

* Paediatric or adult patients with relapsed or refractory CD19+ B cell ALL. (Age 0-60 years). Patients should be in first or subsequent relapse, or relapse after prior stem cell transplant, or persistent Minimal Residual Disease (MRD) positive disease
* ECOG performance score of ≤2 if >16 years old, or Lansky performance score of >50 if ≤16 years old at screening
* Post allogeneic stem cell transplant patients with B cell ALL will be eligible > 3 months after transplant and off immunosuppression for at least 1 month.
* Patients with active leukaemia who developed significant organ impairment that cannot tolerate conventional chemotherapy,
* For women of childbearing potential, a negative pregnancy test prior to apheresis

B-cell lymphoma

* Patients with histologically confirmed refractory Diffuse Large B-cell Lymphoma, primary mediastinal B cell lymphoma or transformed follicular lymphoma or other B-cell lymphoma according to WHO classification
* Confirmed CD19 positivity status in tissue sample obtained at diagnosis or relapse
* Received at least two prior treatment which must include at least one intensive systemic therapy.
* Disease progression or relapsed disease within 12 months after autologous stem cell transplant
* ECOG performance score of ≤2 if >16 years old, or Lansky performance score of >50 if ≤16 years old at screening
* Has sufficient organ function to tolerate treatment with CAR-T cell therapy
* For women of childbearing potential, a negative pregnancy test prior to apheresis

Exclusion criteria of both cohorts

* Patients with active infection
* Patients with B cell ALL post allogeneic transplant with active GVHD or on immunosuppression
* Recent donor lymphocyte infusion (DLI) after allogeneic transplant, less than 6 weeks between DLI and CAR T infusion
* Current autoimmune disease, or history of autoimmune disease with potential CNS involvement
* Active clinically significant CNS dysfunction (including but not limited to uncontrolled seizure disorders, cerebrovascular ischaemia or haemorrhage, dementia, paralysis)
* Patients who are positive for HBsAg, HCV RNA positive or with HIV infection
* Pulmonary function: Grade 1 dyspnea and pulse oxygenation > 91% on room air
* Cardiac function: Fractional shortening <28% or left ventricular ejection fraction <45% by echocardiography.
* Renal function: Creatinine clearance <50 mL/min/1.73 m2
* Liver function: Patients with a serum bilirubin >3 times upper limit of normal or an AST or ALT > 5 times upper limit of normal, unless due to leukaemic liver infiltration in the estimation of the investigator
* Rapidly progressive disease that in the estimation of the investigator would compromise ability to complete study therapy.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Production efficiency of CAR-T cell manufacturing | 18 months
  At least 90% of patients enrolled should be able to achieve successful production of CAR T cells as deomonstrated by CAR-T cell proliferation and persisteance of CAR-T cells in recipients for at least one month after infusion

SECONDARY OUTCOMES:
survival outcome | 24 months
  Achieve a leukemia free survival at 3 months of 60% or higher, and overall survival of B cell ALL patients at 6 months of 50% or higher. Overall and progression free survival of patients with B cell NHL

CONTACTS AND LOCATIONS:
Overall Officials: Chi Kong Li, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
other researchers may approach Principal investigator directly for information